CLINICAL TRIAL: NCT01781715
Title: Multivessel Stenting and Staged Revascularization for ST-elevation Myocardial Infarction Patients With Resolute Integrity Stents
Brief Title: Multivessel Stenting Versus Staged Revascularization With Zotarolimus-eluting Stent for STEMI
Acronym: ZES for STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Vladimir Ganyukov, MD, PhD, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resolute Integrity for STEMI; ZES for STEMI (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: ST Elevation Myocardial Infarction, Multivessel Coronary Artery Disease
Keywords: STEMI, Multivessel Coronary Artery Disease, Primary PCI, multivessel stenting, zotarolimus-eluting stent
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multivessel stenting (Experimental): This group comprises the patients who undergo a one-time primary percutaneous coronary intervention (PCI) of the culprit and nonculprit lesions
  Interventions: Device: Zotarolimus-eluting coronary stent
- Staged revascularization (Active Comparator): This group comprises the patients who undergo PCI of only the culprit lesion and staged nonculprit PCI at a later date (3-15 days)
  Interventions: Device: Zotarolimus-eluting coronary stent

INTERVENTIONS:
Device: Zotarolimus-eluting coronary stent — Multivessel stenting or Staged PCI with Zotarolimus-eluting coronary stent in STEMI patients
  Other Names: Resolute Integrity stent

SUMMARY:
The purpose of this study is to determine outcomes (death, myocardial infarction, target vessel revascularization (TVR), non-target vessel revascularization (non-TVR), stent-thrombosis) of 120 consecutive patients with ST elevation myocardial infarction and multivessel coronary artery disease undergoing multivessel stenting or staged percutaneous coronary intervention with Zotarolimus-eluting stents

DETAILED DESCRIPTION:
Multivessel coronary artery disease has been reported to occur in 40 to 67% of ST elevation myocardial infarction (STEMI) patients. Multivessel coronary artery disease (MVCD) patients, who have experienced STEMI, are at a high risk of major cardiovascular events (MACE) within one year after primary PCI. While MACE incidence in patients with one-vessel coronary artery disease is about 14.5%, patients with two- and three-vessel lesions experience MACE in 19.5% and 23.6% of cases, respectively. The risk of death in a 5-year follow-up increases two-fold in MVCD patients. This risk can be partly explained by slower recovery of left ventricular function and progression of left ventricular pathological remodeling process after MI. In addition, the mere presence of MVCD has been shown to be associated with MACE development in the long-term period. There are several treatment strategies for ST-elevation myocardial infarction (STEMI) patients with MVCD: infarct related artery (IRA)-only percutaneous coronary intervention (PCI), multivessel stenting in the primary PCI setting and staged revascularisation. The current guidelines for STEMI revascularisation give no definite instructions on the need for concurrent non-IRA intervention in patients with stable haemodynamics. At present, there are not clinical trials testing the current Zotarolimus-eluting stents (ZES) in STEMI patients with MVCD undergoing primary PCI for different strategies of revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject is able to verbally confirm understandings of risks, benefits of treatment of either multivessel stenting or staged PCI using the zotarolimus-eluting stent (Resolute Integrity™ Stent, Medtronic) and he or she or his or her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have significant stenoses (≥ 70%) of two or more than two of coronary arteries and requiring primary PCI for acute ST elevation myocardial infarction (STEMI) within 12hrs
* Target lesion(s) must be located in a native coronary artery with visually estimated diameter of less than 2.5 mm and more than 4.0 mm.
* Target lesion(s) must be amenable for percutaneous coronary intervention

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin Aspirin Both Clopidogrel and Ticlopidine, Zotarolimus
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 6 months post enrollment.
* Non-cardiac comorbid conditions are present with life expectancy over 1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Acute heart failure Killip III-IV
* ≥ 50% left main stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
All death including cardiac and non cardiac death | 30 days, 6 months and 12 montrhs
Recurrent MI | 30 days, 6 months and 12 months
Any revascularizations (TLR or TVR) | 30 days, 6 months and 12 months
Composite rate of all death, any MI and any repeat revascularization | 30 days, 6 months and 12 months

SECONDARY OUTCOMES:
stent thrombosis | 30 days. 6 months and 12 months
  The incidence of stent thrombosis was assessed throughout the follow-up period, according to the conventional ARC (Academic Research Consortium) classification.
Non-TVR | 30 days, 6 months and 12 months
  Any repeat revascularization of non target vessels

OTHER OUTCOMES:
Composite rate of all death, any MI and any repeat revascularization | 30 days, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo, Kemerovo Oblast, Russia